CLINICAL TRIAL: NCT01568762
Title: A Randomized, Double-blind, Placebo Controlled Study to Compare the Safety, Tolerability, and Pharmacokinetics of QBX258 (Sequential Administration of a Fixed Dose of VAK694 and Single Ascending Doses of QAX576) in Patients With Well-controlled Mild to Moderate Asthma
Brief Title: To Compare the Safety, Tolerability, and Pharmacokinetics of QBX258 in Patients With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CQBX258X2101
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2012-03

CONDITIONS: Asthma
Keywords: Asthma; VAK694; QAX576; QBX258; pharmacokinetics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- VAK694 (Experimental): VAK694 was administered as a 1 hour intravenous infusion
  Interventions: Drug: VAK694
- VAK694 Placebo (Placebo Comparator): VAK694 placebo was administered as a one hour intravenous infusion
  Interventions: Drug: VAK694 placebo
- QAX576 (Experimental): QAX576 was administered intravenously as a 2 hour infusion
  Interventions: Drug: QAX576
- QAX576 placebo (Placebo Comparator): QAX576 placebo was administered as a 2 hour intravenous infusion
  Interventions: Drug: QAX576 placebo

INTERVENTIONS:
Drug: VAK694 — Intravenous infusion
  Arms: VAK694
Drug: VAK694 placebo — Intravenous infusion
  Arms: VAK694 Placebo
Drug: QAX576 — Intravenous infusion
  Arms: QAX576
Drug: QAX576 placebo — Intravenous infusion
  Arms: QAX576 placebo

SUMMARY:
This study is designed to compare the safety, tolerability, and pharmacokinetics of QBX258 (sequential administration of a fixed dose of VAK694 and single ascending doses of QAX576) in patients with well-controlled mild to moderate asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age 18-60 years (inclusive)
* Well controlled mild to moderate atopic asthma
* Female subjects must be post-menopausal or surgically sterile
* Male subjects must be using two methods of contraception
* Subjects must have a positive skin prick test to one or more common airborne allergen

Exclusion Criteria:

* Participation in any clinical investigation or use of other investigational drugs at time of enrollment
* A history of clinically significant ECG abnormalities
* History of malignancy of any organ system
* Smokers (use of tobacco products in the previous 3 months)
* Use of prescription drugs other than those required for control and relief of asthma
* Use of oral steroids within 12 weeks prior to dosing
* FEVI < 80% predicted at screening or baseline
* Use of albuterol more than twice a week for relief of asthma
* Patients suffering from active hay fever at baseline or likely to require treatment during the study
* History of chronic respiratory disease other than asthma or chronic allergic rhinitis
* Emergency room visit within 6 weeks of screening due to asthma
* Hospitalization for asthma in the last year
* History of intubation/assisted ventilation for asthma in the last 5 years
* Administration of live vaccines within the preceding month

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 100 days
  Adverse events will be determined by evaluating clinical, laboratory evaluations, impact on vital signs and impacts on ECGs

SECONDARY OUTCOMES:
Concentration of serum anti-VAK694 antibodies | Pre-dose, Day 71, 85 and 100
  Blood will be collected to determine concentrations if anti-VAK964 antibodies
Concentration of serum anti-QAX576 antibodies | Pre-dose, Day 71, 85 and 100
  Blood will be collected to determine concentrations if anti-QAX576 antibodies
Area under the serum concentration curve for VAK694 | Pre-dose, 1, 2, 4, 11, 24, 48, 96 hours and Days 8, 15, 29, 43, 57, 71, 85, 100
  Blood will be collected for the measurement of VAK694 serum concentrations
Area under the serum concentration curve for QAX576 | Pre-dose, 1, 2, 4, 11, 24, 48, 96 hours and Days 8, 15, 29, 43, 57, 71, 85, 100
  Blood will be collected for the measurement of QAX576 concentrations
Change in interleukin concentrations | Pre-dose, 1, 2, 4, 11, 24, 48, 96 hours and Days 8, 15, 29, 43, 57, 71, 85, 100
  Blood samples will be collected to measure interleukin concetrations.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Raleigh, North Carolina, United States

REFERENCES:
- See also: Results forCQBX258X2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6763